CLINICAL TRIAL: NCT01262300
Title: Vitamin D Supplementation And Varicella Zoster Virus Vaccine Responsiveness In Older Nursing Home Residents
Brief Title: Vitamin D Supplementation And Varicella Zoster Virus Vaccine Responsiveness In Older Long-Term Care Residents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10-0189; K23AG040708 (NIH)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Immunosenescence; Shingles
Keywords: Immunosenescence; Shingles; Vitamin D; Varicella Zoster Virus; Vaccine; Immune Response; Geriatrics
MeSH Terms: conditions — Herpes Zoster; Chickenpox | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VZV vaccine (Experimental): Varicella Zoster Virus vaccine (Zostavax), single dose X 1 injection
  All subjects in this trial will receive the VZV vaccine. The Investigators will primarily compare immune responses in those that are receiving high dose vs. standard dose vitamin D supplementation and those that have high and low 25-hydroxyvitamin D levels.
  Interventions: Biological: Varicella Zoster Virus Vaccine (Zostavax)

INTERVENTIONS:
Biological: Varicella Zoster Virus Vaccine (Zostavax) — Single 0.65 mL subcutaneous injection of the live, attenuated VZV zoster vaccine (Zostavax; Merck, Whitehouse Station, NJ).

SUMMARY:
This is an ancillary study to a randomized controlled trial of high dose vitamin D in older long-term care residents (NCT01102374). In this study, a subset of trial subjects will receive the zoster vaccine and the investigators will determine the immunological response to the vaccine in this older, frail population, as well as the association between vitamin D and immunological outcomes.

DETAILED DESCRIPTION:
Objectives

1. To determine the increase in Varicella-zoster virus (VZV)-specific cell-mediated immune response from pre-zoster vaccination to 3 weeks post-vaccination in nursing home residents after 4 months of high dose vs. standard dose vitamin D3 supplementation.
2. In the same participants as Aim 1, to measure the association between pre-zoster vaccination 25-hydroxyvitamin D [25(OH)D] levels and the increase in VZV-specific cell-mediated immune response from pre- vaccination to 3 weeks post-vaccination.
3. Characterize the phenotypic and functional VZV-specific T cell responses to Zostavax, including memory, effector, Th1/Th2, and homing receptor-bearing T cells in the high compared to low ELISPOT responders.

Hypotheses

1. At baseline, higher serum 25(OH)D levels will be associated with higher levels of VZV-specific cell-mediated immunity (cross-sectional).
2. At baseline, higher serum 25(OH)D levels, independent of vitamin D supplementation dose, will be associated with greater increases in VZV-specific cell-mediated immune responses to Zostavax, as measured by the interferon (IFN)-γ ELISPOT assay.
3. Compared to standard dose, high dose vitamin D3 supplementation will enhance VZV-specific cell-mediated immune response to vaccination independent of baseline serum 25(OH)D levels.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 60 years;
2. Residing in a long-term care facility;
3. Have not yet received VZV vaccine

Exclusion Criteria:

1. terminal illness (expected survival <6 months);
2. anticipated discharge within 12 months;
3. unable to take whole or crushed tablets;
4. active cancer, except squamous/basal cell carcinoma;
5. severe malnutrition (body mass index <18 kg/m2);
6. current immunosuppressive medications (including corticosteroids);
7. renal failure (eGFR<15 mL/min/1.73m2);
8. currently taking >800 IU/d vitamin D supplementation;
9. history (or strong family history) of kidney stones;
10. history of sarcoidosis or other granulomatous disorders associated with hypercalcemia;
11. elevated baseline hypercalcemia (albumin-adjusted serum calcium >10.5 mg/dL);
12. serum 25 (OH)D level ≥40 ngl/ml at baseline;
13. inability to provide informed consent and no available healthcare proxy;
14. inability of participant or proxy to speak/understand English.
15. previous receipt of the Zostavax (anticipate <10% of trial;
16. known allergy to gelatin, neomycin, or any other component of the vaccine.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01-23 (Actual); Study Completion 2014-01-23 (Actual)

PRIMARY OUTCOMES:
VZV-specific cell mediated immunity, as measured by the interferon-γ ELISPOT assay | 3 weeks post-vaccination

SECONDARY OUTCOMES:
VZV-gpELISA to measure the VZV-specific antibody concentration | 3 weeks post-vaccination
VZV-specific effector and memory T cells | 3 weeks post-vaccination
-specific cell mediated immunity, as measured by the responder cell frequency assay | 3 weeks post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Adit A Ginde, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] A randomized controlled trial of high dose vitamin D in older long-term care residents (NCT01102374)